CLINICAL TRIAL: NCT02239705
Title: Mathematical Coupling of Data Between Global-End Diastolic Volume Index and Cardiac Index Calculated by Edwards EV1000
Brief Title: Mathematical Coupling of Data in Transpulmonary Thermodilution
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Alberto Sciusco, Medical doctor, University of Foggia
Other Study IDs: A02
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Critical Illness
Keywords: Trans pulmonary thermodilution; Hemodynamic
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fluid challenge: Patients whose clinical conditions require bolus of fluids infusion to correct blood pressure and cardiac output
- Inotropic infusion: Patient whose clinical conditions require inotropic agents infusion to correct blood pressure and cardiac output

SUMMARY:
The purpose of this study is to investigate whether cardiac output (CO) and global end diastolic volume (GEDV) determined from the same thermodilution curve by EV1000 are mathematically coupled during the infusion of fluid or inotropic agents in critically ill patients.

DETAILED DESCRIPTION:
Some fundamental questions remain unanswered about the mathematical analysis of the thermodilution curve and the physiological significance of the Global End Diastolic Volume ( GEDV ) .

The mathematical derivation of the Global End Diastolic Volume (GEDV) is intimately linked with the Cardiac Output (CO), because EV1000, to calculate the GEDV, uses a formula in which the CO is the term "flow " for both the calculations of Volume Thermal Intra Thoracic (ITTV) and Lung Thermal volume (PTV) .

The clinical validation of GEDV as an index of preload has been substantially based on measuring changes in GEDV and CO in response to the Fluid Challenge only in patients "volume responsive".

In this scenario, GEDV and CO may show a close correlation only on the basis of their mathematical derivation.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted in the Intensive Care Department
* patient monitored by EV1000 trans pulmonary device
* Systolic blood pressure (SBP) less than 90 mm Hg or SBP Drop ≥ 40 mm Hg of normal
* decision by 1 expert intensivist physician to initiate fluid resuscitation hospital protocol or therapeutic infusion of vasopressor agent

Exclusion Criteria:

* pregnancy
* age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiac Output | Triplicate measurement in each subject before and 20 minutes after therapeutic infusion of fluids or vasopressor agents
  To evaluate the change in cardiac function after therapeutic life-saving fluid resuscitation or vasopressor agent infusion, cardiac output will be assessed before and after 20 minutes starting infusion.
Change in Global end diastolic volume | Triplicate measurement in each subject before and 20 minutes after therapeutic infusion of fluids or vasopressor agents
  To evaluate the change in cardiac function after therapeutic life-saving fluid resuscitation or vasopressor agent infusion, global end diastolic volume will be assessed before and after 20 minutes starting infusion.
Change Left ventricular volume | Before and 20 minutes after therapeutic infusion of fluids or vasopressor agents
  To evaluate the change in cardiac function after therapeutic, life-saving fluid resuscitation or vasopressor agent infusion, Left ventricular volume measurement with echocardiography will be evaluated before and after 20 minutes starting infusion.
Change Right ventricular volume | Before and 20 minutes after therapeutic infusion of fluids or vasopressor agents
  To evaluate the change in cardiac function after therapeutic life-saving fluid resuscitation or vasopressor agent infusion, Right Ventricular Volume measurement with echocardiography will be assessed before and after 20 minutes starting infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Dambrosio, Medic, Study Chair — University of Foggia; Livio Tullo, Medic, Study Director — University of Foggia; Alberto Sciusco, medic, Principal Investigator — University of Foggia
Locations (1):
- Ospedali Riuniti, Foggia, FG, Italy

REFERENCES:
- See also: Speciality school of anesthesia of University of Foggia — http://www.anestesia.unifg.it/Segreteria-e-Contatti/179/